CLINICAL TRIAL: NCT01209117
Title: A Single-center, Randomized, Open-label, Crossover Study to Assess the Relative Bioavailability of Tablet Formulations of GSK2248761 in Healthy Adult Subjects. SGN114435
Brief Title: A Study to Assess the Relative Bioavailability of Tablet Formulations of GSK2248761 in Healthy Adult Subjects. SGN114435
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 114435
Record Dates: First submitted 2010-09-17; First posted 2010-09-27 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Infections, Human Immunodeficiency Virus and Herpesviridae; Infection, Human Immunodeficiency Virus
Keywords: formulation; bioavailability; pharmacokinetics; GSK2248761
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Periods 1 - 4 (Experimental): Subjects will be randomized in a cross over fashion to receive the GSK2248761 WBM capsule formulation or one of three WBM tablet formulations in one of four sequences.
  Interventions: Drug: GSK2248761 WBM Capsule; Drug: GSK2248761 WBM Tablet Formulation 1; Drug: GSK2248761 WBM Tablet Formulation 2; Drug: GSK2248761 WBM Tablet Formulation 3
- Period 5 (Experimental): Subjects in Part B will receive a formulation of GSK2248761 200mg WBM Tablet chosen from Periods 1 - 4 in part A in the fed state (moderate fat meal).
  Interventions: Drug: GSK2248761 WBM Tablet

INTERVENTIONS:
Drug: GSK2248761 WBM Capsule — 200 mg GSK2248761 WBM capsule (reference) 2 X100mg
  Arms: Periods 1 - 4
Drug: GSK2248761 WBM Tablet Formulation 1 — GSK2248761 WBM Tablet 200mg manufacturing process 1
  Arms: Periods 1 - 4
Drug: GSK2248761 WBM Tablet Formulation 2 — GSK2248761 WBM Tablet 200mg manufacturing process 2
  Arms: Periods 1 - 4
Drug: GSK2248761 WBM Tablet Formulation 3 — GSK2248761 WBM Tablet 200mg manufacturing process 3
  Arms: Periods 1 - 4
Drug: GSK2248761 WBM Tablet — GSK2248761 WBM tablet 200mg manufacturing process 1, 2, or 3 chosen from Period 1 - 4
  Arms: Period 5

SUMMARY:
This is a single-center, randomized, two part, open-label, crossover study in healthy adult subjects to assess the oral bioavailability of three GSK2248761 Wet Bead Milled (WBM) tablet formulations manufactured by three different processes relative to the GSK2248761 WBM capsule formulation (Part A) and the effect of a moderate-fat meal on the bioavailability of the selected WBM tablet formulation (Part B).

DETAILED DESCRIPTION:
ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, vital signs, laboratory tests, and ECGs. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 50 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any female who: Is pre-menopausal with a documented bilateral tubal ligation, bilateral oophorectomy (removal of the ovaries) or hysterectomy, or Is post-menopausal defined as 12 months of spontaneous amenorrhea.
* Male subjects must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until the follow-up visit.
* Body weight greater than or equal to 50 kilograms (kg) for men and greater than or equal to 45 kg for women and body mass index (BMI) within the range 18.5-31.0 kilograms per meters squared (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* As a result of the medical interview, physical examination, or screening investigations, the Investigator considers the subject unfit for the study.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* Unwilling to refrain from the use of illicit drugs and adhere to other protocol-stated restrictions while participating in the study.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of greater than14 drinks/week for men or greater than 7 drinks/week for women.
* Unwilling to abstain from alcohol for 48 hours prior to the start of dosing until collection of the final pharmacokinetic sample during each treatment period.
* History or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting surgery or percutaneous transluminal coronary angioplasty or any clinically significant cardiac disease.
* History/evidence of clinically significant pulmonary disease.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy should be excluded.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* Where participation in the study would result in donation of blood or blood products in excess of 500 milliliters (mL) within a 56 day period.

Note: this does not include plasma donation.

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* aspartate aminotransferase (AST), alanine aminotransferase (ALT) , alkaline phosphatase and bilirubin greater than or equal to 1.5 times the Upper limit of normal (isolated bilirubin >1.5 times the upper limit of normal is acceptable if bilirubin is fractionated and direct bilirubin less than 35%).
* Pregnant females as determined by positive serum pregnancy test at screening or prior to dosing.
* Lactating females.
* The subject's systolic blood pressure is outside the range of 90-140 millimeters of mercury, or diastolic blood pressure is outside the range of 45-90millimeters of mercury or heart rate is outside the range of 50-100beats per minute for female subjects or 45-100 beats per minute for male subjects at Screening and predose Day 1.
* Cardiac conduction abnormalities denoted by any of the following on a single 12-lead ECG at screening or predose Day 1.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Plasma GSK2248761 Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC(0-infinity)) | 5 weeks
Plasma GSK2248761 Area under the concentration-time curve over the dosing interval (AUC (0 - t)) | 5 weeks
Plasma GSK2248761 observed concentration 24 hours after dose (C24) | 5 weeks
Plasma GSK2248761 Maximum observed concentration (Cmax) | 5 weeks

SECONDARY OUTCOMES:
Safety and tolerability parameters, including adverse events | 5 weeks
concurrent medication | 5 weeks
Clinical laboratory screens | 5 weeks
Electrocardiograms (ECG) | 5 weeks
Vital sign assessments (systolic and diastolic blood pressure and pulse) | 5 weeks
Plasma GSK2248761 terminal phase half life (t½) | 5 weeks
Plasma GSK2248761 Lag time before observation of drug concentrations (tlag) | 5 weeks
Plasma GSK2248761 Time of occurrence of Cmax (tmax) | 5 weeks
Plasma GSK2248761 Percentage of AUC(0-infinity) obtained by extrapolation (%AUCex) | 5 weeks
Plasma GSK2248761 Time of last quantifiable concentration (tlast) | 5 weeks
Plasma GSK2248761 Apparent clearance following oral dosing (CL/F) | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States